CLINICAL TRIAL: NCT01740531
Title: A Randomized Controlled Study to Evaluate Efficacy and Safety of S 303 Treated Red Blood Cells (RBC) in Subjects With Thalassemia Major Requiring Chronic RBC Transfusion
Brief Title: Study to Evaluate Efficacy and Safety of S303 Treated Red Blood Cells (RBCs)in Subjects With Thalassemia Major Requiring Chronic RBC Transfusion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CLI 00076
Record Dates: First submitted 2012-11-21; First posted 2012-12-04 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Thalassemia Major
Keywords: S303 treated RBCs
MeSH Terms: conditions — beta-Thalassemia | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-303 Treated Red Blood Cells (RBC) (Experimental): Patients will be randomly assigned to the sequence of administration of Test and Control RBCs; eligible patients are randomly assigned to receive Test RBCs followed by Control RBCs or Control RBCs followed by Test RBCs. Each patient will complete both treatment periods.
  Interventions: Biological: S-303 Treated Red Blood Cells (RBCs)
- Conventional, untreated Red Blood Cells (Active Comparator): Patients will be randomly assigned to the sequence of administration of Test and Control RBCs; eligible patients are randomly assigned to receive Test RBCs followed by Control RBCs or Control RBCs followed by Test RBCs. Each patient will complete both treatment periods.
  Interventions: Biological: Conventional, untreated Red Blood Cells

INTERVENTIONS:
Biological: S-303 Treated Red Blood Cells (RBCs)
  Arms: S-303 Treated Red Blood Cells (RBC)
Biological: Conventional, untreated Red Blood Cells
  Arms: Conventional, untreated Red Blood Cells

SUMMARY:
To evaluate the efficacy and safety of S 303 treated red blood cells (RBCs) in subjects who require chronic transfusion support due to thalassemia major.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of S 303 treated red blood cells (RBCs) in subjects who require chronic transfusion support due to thalassemia major.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥10 years, of either gender
* Diagnosed with thalassemia major and currently participating in a chronic transfusion program
* At least a one year history of chronic RBC transfusion support with a stable transfusion requirement (per treating physician)
* Intervals of at least 14 days between RBC transfusions
* All RBC components are given on one day for each transfusion episode
* Negative direct antiglobulin tests (DAT)
* Stable iron chelation regimen
* Available for measurement of hemoglobin level at one hour post transfusion
* Signed and dated informed consent form

Exclusion Criteria:

* Baseline antibody specific to S 303 treated RBC (positive test, as defined in Section 8.4.1)
* Evidence of splenic hyper function defined as a transfusion requirement >180 cc/kg/year (at 100% hematocrit)
* Splenic enlargement: spleen palpable ≥4 cm below costal margin OR ≥18 cm in longitudinal diameter by ultrasound (chosen at the Investigator's discretion according to the data available with ultrasound data being preferable)
* Any subject for whom a transition in the number of RBC units transfused is anticipated within 12 months of study entry due to growth of the subject (e.g. a transition from 1 RBC component per transfusion cycle to 2 OR a transition from 2 to 3 is anticipated based on weight change alone)
* Alloimmunization to high frequency blood group antigens to the extent that the ready provision of compatible blood may not be feasible for the study (alloimmunization alone is not an automatic exclusion)
* Current specialized treatment with washed or frozen RBC
* Requirement for gamma irradiated RBC components (would present blinding difficulty due to blood component labeling regulations
* Treatment with any medication that is known to adversely affect RBC viability
* HIV infection (defined as RNA positive)
* HCV (hepatitis C)infection (defined as RNA positive) if treated with concomitant medications known to suppress the bone marrow
* Pregnant or breast feeding female, or female of child bearing potential not using a medically approved form of contraception
* Acute or chronic medical disorder other than thalassemia that, in the opinion of the Investigator or medical monitor, may prevent the subject from completing participation in the study
* Participation in another clinical study, either concurrently or within the previous 28 days, in which the study drug or device may influence red blood cell viability

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint - Hemoglobin consumption | 12 months
  Hemoglobin consumption measured as total hemoglobin mass transfused per subject adjusted for average body weight and the number of days during the efficacy evaluation period (adjusted hemoglobin (Hgb) consumption units are g Hgb/kg body weight/day).
Primary Safety Endpoint-Incidence of a treatment-emergent antibody with confirmed specificity to S 303 treated red blood cells (RBC) | 12 months
  Incidence of a treatment-emergent antibody with confirmed specificity to S 303 treated red blood cells (RBC) associated with clinically significant hemolysis

SECONDARY OUTCOMES:
Secondary Efficacy Endpoint-Hemoglobin increment | 12 months
  Hemoglobin increment one hour post-transfusion
Secondary Efficacy Endpoint-Proportional decline in post transfusion hemoglobin level per day (%/day) | 12 months
  Proportional decline in post transfusion hemoglobin level per day (%/day)
Secondary Safety Endpoint-Adverse Events | 12 months
  Subjects will be actively monitored for adverse events during the transfusion episode and until discharge from the transfusion clinic.
Secondary Safety Endpoint-Transfusion reactions within 24 hours | 12 Months
  Transfusion reactions within 24 hours of a study transfusion with the assigned study product.
Secondary Safety Endpoint-Frequency of allo immunization to red blood cell (RBC) allo-antigens | 12 months
  Frequency of allo immunization to red blood cell (RBC) allo-antigens

CONTACTS AND LOCATIONS:
Overall Officials: Raffaella Origa, MD, Principal Investigator — Ospedale Regionale per le Microcitemie azienda; Antonio Piga, MD, Principal Investigator — University of Torino; Yesim Aydinok, MD, Principal Investigator — Ege University, Izmir, Turkey
Locations (3):
- Italy (2):
  - Ospedale Regionale per le Microcitemie Azienda, Cagliari
  - University of Torino, Torino
- Ege University, Izmir, Turkey (Türkiye)